CLINICAL TRIAL: NCT03433092
Title: Serum Carotenoids and Risk of Gastrointestinal Tract Cancer: Meta-analysis of Ten Studies
Status: Completed | Type: Observational
Sponsor: Yong Zhou (Other)
Collaborators: Sichuan Provincial Science and Technology Support Project (2016SZ0047) (Unknown)
Responsible Party: Sponsor-Investigator, Yong Zhou, West China Hospital, West China Hospital
Organization: West China Hospital (Other)
Other Study IDs: 2759067085
Record Dates: First submitted 2018-02-07; First posted 2018-02-14 (Actual); Last update posted 2018-02-22 (Actual); Status verified 2018-02

CONDITIONS: Gastrointestinal Tract Cancer
Keywords: Serum carotenoids; Gastrointestinal tract cancer; Meta-analysis
MeSH Terms: conditions — Gastrointestinal Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (10):
- Jing Huang et. al, 2017
  Interventions: Other: serum carotenoids
- Max Leenders et. al,2014
  Interventions: Other: serum carotenoids
- Yusuke Okuyama et. al,2014
  Interventions: Other: serum carotenoids
- GC Kabat et. al,2012
  Interventions: Other: serum carotenoids
- Christina Persson et. al,2008
  Interventions: Other: serum carotenoids
- M Jenab et. al,2006
  Interventions: Other: serum carotenoids
- Kenji Wakai et. al,2005
  Interventions: Other: serum carotenoids
- Christian C. Abnet et. al,2003
  Interventions: Other: serum carotenoids
- N Malila et. al,2002
  Interventions: Other: serum carotenoids
- G Pappalardo et. al,1997
  Interventions: Other: serum carotenoids

INTERVENTIONS:
Other: serum carotenoids — In each study, the serum concentrations of carotenoids were detected by high performance liquid chromatography

SUMMARY:
Previous studies have suggested that serum carotenoids may be associated with risk of gastrointestinal tract cancer (GIT cancer), but the results were inconsistent. Thus, the investigators conducted a meta-analysis to evaluate the associations between serum carotenoids and risk of GIT cancer.

ELIGIBILITY:
Inclusion Criteria:

* The study had both case and control groups
* Serum carotenoids levels, relative risk (RR) or OR and corresponding 95% CI were reported
* Patients in case group were diagnosed with GIT cancer

Exclusion Criteria:

·Animal studies

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: The study population include people from primary care clinic or community sample.
Sampling Method: Probability Sample
Enrollment: 40641 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2017-11-20 (Actual); Study Completion 2017-12-28 (Actual)

PRIMARY OUTCOMES:
Gastrointestinal Tract Cancer Incident Measure | Through study completion, an average of 5 years.
  The gastrointestinal tract cancer incident would be recorded during the follow-up years.

CONTACTS AND LOCATIONS:
Locations (1):
- West China Hospital, Sichuan University, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Huang J, Lu MS, Fang YJ, Xu M, Huang WQ, Pan ZZ, Chen YM, Zhang CX. Serum carotenoids and colorectal cancer risk: A case-control study in Guangdong, China. Mol Nutr Food Res. 2017 Oct;61(10). doi: 10.1002/mnfr.201700267. Epub 2017 Jul 31. PMID 28605127